CLINICAL TRIAL: NCT02713490
Title: A Multicenter, Randomized, Double-Blind, Controlled Trial Comparing Local Infiltration Analgesia With EXPAREL to Local Infiltration Analgesia Without EXPAREL to Manage Postsurgical Pain Following Total Knee Arthroplasty
Brief Title: Local Infiltration Analgesia With and Without EXPAREL Following Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 402-C-331
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EXPAREL (Active Comparator): Single dose of EXPAREL 266 mg in 20 mL admixed with bupivacaine HCl 0.5% in 20 mL and expanded in volume with 80 mL normal saline (total volume of 120 mL).
  Interventions: Drug: EXPAREL
- Bupivacaine (Active Comparator): Bupivacaine HCl 0.5% in 20 mL expanded in volume with 100 mL normal saline (total volume of 120 mL).
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: EXPAREL — EXPAREL and bupivacaine HCl
  Other Names: bupivacaine liposome injectable suspension
  Arms: EXPAREL
Drug: Bupivacaine — Single dose of bupivacaine HCl 0.5%
  Other Names: bupivacaine HCl
  Arms: Bupivacaine

SUMMARY:
This is a Phase 4, multicenter, randomized, double-blind, controlled trial in approximately 140 adult subjects undergoing primary unilateral TKA under spinal anesthesia with bupivacaine HCl (10-15 mg).

DETAILED DESCRIPTION:
On Day 0, eligible subjects will be randomized 1:1 to two treatment groups. Subjects in Group 1 will receive local infiltration analgesia (LIA) with EXPAREL 266 mg in 20 mL admixed with bupivacaine hydrochloride (HCl) 0.5% in 20 mL and expanded in volume with 80 mL normal saline (total volume of 120 mL). Subjects in Group 2 will receive LIA with bupivacaine HCl 0.5% in 20 mL expanded in volume with 100 mL normal saline (total volume of 120 mL). Investigators will use their usual surgical technique to perform the TKA.

Study drug will be administered using six 20 cc syringes with 22-gauge needles prior to wound closure. Each stick should deliver approximately 1-1.5 cc to the intended area. The tissue should visibly expand with minimal leakage. Study drug should be injected in the prescribed locations based on the areas of highest nerve density.

Infiltration Technique

Prior to cementation

Syringe #1: Posterior capsule (8-10 sticks medial and 8-10 sticks lateral).

Syringe #2: Femur medial and lateral periosteum, posterior periosteum, suprapatellar/quadriceps tendon (20 sticks).

Syringe #3: Tibia fat pad (5 sticks); pes anserinus, medial collateral ligament, and gutter (15 sticks).

Syringe #4: Circumferential periosteum (15-20 sticks).

After cementation

Syringe #5: Midline quadriceps tendon (10 sticks); retinaculum, medial gutter, femoral to tibia (10 sticks).

Syringe #6: Lateral gutter, femoral to tibial (10 sticks); subcutaneous/closure (10 sticks).

In addition to LIA, all study participants will receive a standardized approach for managing postsurgical pain that includes a scheduled multimodal pain regimen including adjunctive analgesics, non-steroidal anti-inflammatory drugs (NSAIDs), and rescue analgesics as needed.

Postsurgical clinical assessments will include pain intensity scores using a 10-cm visual analog scale (VAS); overall benefit of analgesia score (OBAS) questionnaire; total postsurgical opioid consumption; physical therapy assessment; nurse's satisfaction with overall analgesia; and discharge readiness. Adverse events (AEs) will be recorded from the time the informed consent form is signed through postsurgical Day 29.

Postsurgical health economic outcome assessments will include hospital length of stay (LOS), use of skilled nursing facility, outpatient physical therapy use, hospital readmissions, and use of other health services following discharge (phone calls related to postsurgical pain, unscheduled visits related to postsurgical pain, and visits to emergency department) through postsurgical Day 29.

A follow-up visit will be scheduled for all subjects on postsurgical Day 14. A follow-up phone call will be made on postsurgical Day 29 to all subjects who received study drug to assess for AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age at screening.
2. Scheduled to undergo primary, unilateral, tricompartmental TKA under spinal anesthesia.
3. Primary indication for TKA is degenerative osteoarthritis of the knee.
4. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.
5. Female subjects must be surgically sterile; or at least 2 years postmenopausal; or have a monogamous partner who is surgically sterile; or practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than 2 months prior to screening and commit to the use of an acceptable form of birth control for the duration of the study and for 30 days after completion of the study.
6. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration.
2. History of previous prior contralateral TKA or open knee surgery on the knee being considered for TKA. Prior arthroscopy is permitted.
3. Planned concurrent surgical procedure (e.g., bilateral TKA).
4. Undergoing unicompartmental TKA or revision TKA.
5. Concurrent painful physical condition that may require analgesic treatment (such as an NSAID or opioid) in the postsurgical period for pain that is not strictly related to the knee surgery and which may confound the postsurgical assessments (e.g., significant pain from other joints including the non-index knee joint, chronic neuropathic pain, concurrent or prior contralateral TKA, concurrent foot surgery).
6. Comorbidity impacting current physical function of Investigator opinion that it may impact postsurgical rehabilitation.
7. Allergy, hypersensitivity, or contraindication to any of the study medications (i.e., bupivacaine, pregabalin, acetaminophen/paracetamol, celecoxib, oxycodone, morphine, hydromorphone, or tranexamic acid).
8. Use of any of the following medications within the times specified before surgery: long-acting opioid medication or NSAIDs (except for low-dose aspirin used for cardioprotection) within 3 days, or any opioid medication within 24 hours.
9. Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®). If a subject is taking one of these medications for a reason other than pain control, he or she must be on a stable dose for at least 1 month prior to study drug administration.
10. Current use of systemic glucocorticosteroids within 1 month of enrollment in this study.
11. Use of dexmedetomidine HCl (Precedex®) within 3 days of study drug administration.
12. History of coronary or vascular stent placed within the past 3 months (may be extended to 1 year if medically indicated per physician discretion).
13. Have been treated for a deep vein thrombosis, pulmonary embolism, myocardial infarction, or ischemic stroke within the past 6 months (may be extended to 1 year if medically indicated per physician discretion).
14. Rheumatoid or inflammatory arthritis or disease.
15. Severely impaired renal or hepatic function (e.g., serum creatinine level >2 mg/dL [176.8 µmol/L], blood urea nitrogen level >50 mg/dL [17.9 mmol/L], serum aspartate aminotransferase [AST] level >3 times the upper limit of normal [ULN], or serum alanine aminotransferase [ALT] level >3 times the ULN.)
16. Any neurologic or psychiatric disorder that might impact postsurgical pain or interfere with study assessments.
17. Malignancy in the last 2 years, per physician discretion.
18. History of misuse, abuse, or dependence on opioid analgesics, other prescription drugs, illicit drugs, or alcohol.
19. Failure to pass the alcohol breath test or urine drug screen.
20. Body weight <50 kg (110 pounds) or a body mass index >40 kg/m2.
21. Previous participation in an EXPAREL study.
22. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-04-18; Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Jones, MD, PharmD, Study Director — Pacira Pharmaceuticals, Inc
Locations (17):
- United States (17):
  - Institute for Joint Restoration, Fremont, California
  - Loma Linda University, Loma Linda, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Pinnacle Orthopaedics & Sports, Marietta, Georgia
  - Central DuPage Hospital, Northwestern Medicine, Winfield, Illinois
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Orthopaedic Associates, Towson, Maryland
  - NYU Hospital for Joint Disease, New York, New York
  - Lenox Hill Hospital/Northwell Health Orthopaedic Institute, New York, New York
  - UNC Orthopaedics Chapel Hill, Chapel Hill, North Carolina
  - OrthoCarolina, PA, Charlotte, North Carolina
  - Wellington Orthopaedics and Sports Medicine, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Baylor Medical Center, Plano Orthopedics Sports Medical & Spine Center, Frisco, Texas
  - Utah University Orthopedic Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dysart SH, Barrington JW, Del Gaizo DJ, Sodhi N, Mont MA. Local Infiltration Analgesia With Liposomal Bupivacaine Improves Early Outcomes After Total Knee Arthroplasty: 24-Hour Data From the PILLAR Study. J Arthroplasty. 2019 May;34(5):882-886.e1. doi: 10.1016/j.arth.2018.12.026. Epub 2018 Dec 25. PMID 30799269
- [Derived] Mont MA, Beaver WB, Dysart SH, Barrington JW, Del Gaizo DJ. Local Infiltration Analgesia With Liposomal Bupivacaine Improves Pain Scores and Reduces Opioid Use After Total Knee Arthroplasty: Results of a Randomized Controlled Trial. J Arthroplasty. 2018 Jan;33(1):90-96. doi: 10.1016/j.arth.2017.07.024. Epub 2017 Jul 25. PMID 28802777

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between April 18, 2016 and February 8, 2017 at 16 sites in the United States
Pre-assignment Details: A total of 167 patients were screened; there were 27 screen failures, including 2 patients who were randomized in error to the EXPAREL 266 mg + bupivacaine hydrochloride (HCl) group.
Groups:
- EXPAREL 266 mg + Bupivacaine HCl: Local infiltration analgesia with EXPAREL (bupivacaine liposome injectable suspension) 266 mg/20 mL admixed with bupivacaine HCl 0.5% 20 mL and expanded with 80 mL normal saline
- Bupivacaine HCl: Local infiltration analgesia with bupivacaine HCl 0.5% 20 mL expanded with 100 mL normal saline
Period: Overall Study
Arm/Group | EXPAREL 266 mg + Bupivacaine HCl | Bupivacaine HCl
Started | 71 | 69
Completed | 68 | 67
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Did not receive study drug | 1 | 0
Not completed — Met exclusion criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received study drug, with analysis by actual treatment received.
Groups:
- EXPAREL: Local infiltration analgesia with EXPAREL (bupivacaine liposome injectable suspension) 266 mg/20 mL admixed with bupivacaine HCl 0.5% 20 mL and expanded with 80 mL normal saline
- Bupivacaine: Local infiltration analgesia with bupivacaine HCl 0.5% 20 mL expanded with 100 mL normal saline
- Total: Total of all reporting groups
Arm/Group | EXPAREL | Bupivacaine | Total
Number analyzed (Participants) | 70 | 69 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (8.61) | 65.8 (7.21) | 65.8 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 27 | 30 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 66 | 68 | 134
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 61 | 61 | 122
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 70 | 69 | 139
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.395 (5.805) | 31.311 (5.189) | 31.857 (5.515)
VAS pain score [Mean (Standard Deviation); unit: cm] — Visual Analog Scale (VAS) is a pain scale. The VAS was presented as a straight 10 cm line, where 0 cm is no pain and 10 cm is the worst pain possible. Patients were asked, "How much pain are you experiencing right now? Please place a vertical mark on the line below to indicate the level of pain you are experiencing right now." Population: Two patients in the EXPAREL 266 mg + bupivacaine HCl group did not have VAS measurements entered in the database.
  cm
    number analyzed (Participants) | 68 | 69 | 137
    (all) | 1.91 (2.120) | 1.89 (2.241) | 1.90 (2.174)
American Association of Anesthesiologists classification [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) classification was determined by physicians using the ASA Physical Status Classification System which assesses the patient's pre-anesthesia medical co-morbidities. ASA 1 patients would be considered a normal, healthy patient. ASA 2 is a patient with mild systemic disease (eg, smoker, well controlled diabetes or high blood pressure (HBP)). ASA 3 is a patient with severe systemic disease (eg poorly controlled diabetes or HBP). ASA 4 is a patient with severe systemic disease that is a constant threat to life (eg, recent myocardial infarction, stroke).
  Participants
    1 | 3 | 2 | 5
    2 | 45 | 40 | 85
    3 | 22 | 27 | 49
Location of surgery [Count of Participants; unit: Participants]
  Left | 31 | 25 | 56
  Right | 39 | 44 | 83

OUTCOME MEASURES:

1. Primary Outcome: Area Under The Curve (AUC) of Visual Analog Scale (VAS) Pain Intensity Scores From 12 to 48 Hours
Description: AUC of VAS pain intensity scores from 12 to 48 hours, which represents total pain experienced from 12 to 48 hours. Visual Analog Scale (VAS) is a pain scale. The VAS was presented as a straight 10 cm line, where 0 cm is no pain and 10 cm is the worst pain possible. Patients were asked, "How much pain are you experiencing right now? Please place a vertical mark on the line below to indicate the level of pain you are experiencing right now."
Time Frame: From 12-48 hours
Population: Efficacy population: all participants who received study drug and underwent the surgery, with analysis based on randomized treatment
Measure: Least Squares Mean (Standard Error); unit: cm*hr
Arm/Group | EXPAREL | Bupivacaine
Number analyzed (Participants) | 69 | 69
cm*hr | 181.523 (10.786) | 208.407 (10.814)
Statistical Analysis 1: Comparison: EXPAREL vs Bupivacaine; Test type: Superiority; p = 0.0381, ANOVA; LSMD = -26.884, 95% CI 2-sided [-56.608 to 2.841]

2. Primary Outcome: Total Postsurgical Opioid Consumption Through 48 Hours
Description: Total postsurgical opioid consumption (converted to oral morphine equivalents) through 48 hours
Time Frame: 0-48 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | EXPAREL | Bupivacaine
Number analyzed (Participants) | 70 | 69
mg | 16.321 (6.684) | 80.328 (33.249)
Statistical Analysis 1: Comparison: EXPAREL vs Bupivacaine; Test type: Superiority; p = 0.0029, ANOVA; LSM treatment ratio = 0.203, 95% CI 2-sided [0.065 to 0.631]

3. Secondary Outcome: Percentage of Opioid-free Subjects at 48 Hours
Time Frame: 48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EXPAREL | Bupivacaine
Number analyzed (Participants) | 70 | 69
Participants | 7 | 0
Statistical Analysis 1: Comparison: EXPAREL vs Bupivacaine; Test type: Superiority; p = 0.0088, Cochran-Mantel-Haenszel; Treatment difference = 0.098, 95% CI 2-sided [0.0284 to 0.1685]

4. Secondary Outcome: Time to First Opioid Rescue in the First 48 Hours
Description: Time to first opioid rescue was estimated from Kaplan-Meier analysis and presented as quartiles (ie, time to rescue for the first 25% / 50% / 75% of subjects within each treatment group).
Time Frame: 48 hours
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: h
Arm/Group | EXPAREL | Bupivacaine
Number analyzed (Participants) | 70 | 69
h
  First quartile | 2.617 [1.083 to 3.233] | 1.00 [0.600 to 1.967]
  Median quartile | 4.125 [3.333 to 6.133] | 2.917 [2.083 to 3.883]
  Third quartile | 9.667 [6.250 to 31.083] | 7.200 [4.00 to 12.600]
Statistical Analysis 1: Comparison: EXPAREL vs Bupivacaine; Analysis applies to the overall distribution of time to first opioid rescue, estimated from Kaplan-Meier analysis; Test type: Superiority; p = 0.0230, Log Rank

5. Secondary Outcome: Overall Benefit of Analgesia Score at 48 Hours
Description: The overall benefit of analgesic score (OBAS) comprises seven questions to assess pain intensity, adverse effects, and patients' satisfaction with analgesia (eg, "Please rate your current pain at rest on a scale between 0=minimal pain and 4=maximum imaginable pain"). Overall scores ranged between 0- 28. OBAS measures patients' benefit from postoperative pain therapy. A lower composite score indicates greater benefit from the therapy.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EXPAREL | Bupivacaine
Number analyzed (Participants) | 70 | 69
score on a scale | 4.1 (4.08) | 4.6 (4.33)
Statistical Analysis 1: Comparison: EXPAREL vs Bupivacaine; Test type: Superiority; p = 0.4285, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: From screening to postsurgical day 29
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (eg, abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug without any judgment about causality. Serious AEs were defined as per clinicaltrials.gov.
  Note that 71 subjects were randomized into the EXPAREL arm, but only 70 subjects received EXPAREL.
Arm/Group | EXPAREL | Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 1/70 | 1/69
Other Adverse Events (participants affected / at risk) | 45/70 | 39/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL (N=70) | Bupivacaine (N=69)
Incision site cellulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL (N=70) | Bupivacaine (N=69)
Nausea (Gastrointestinal disorders) | 21 | 22
Anemia (Blood and lymphatic system disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 3 | 3
Peripheral swelling (General disorders) | 1 | 3
Hypotension (Vascular disorders) | 3 | 1
Anemia postoperative (Injury, poisoning and procedural complications) | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 3 | 8
Insomnia (Psychiatric disorders) | 3 | 2
Mental status change (Psychiatric disorders) | 0 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 0
Bradycardia (Cardiac disorders) | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Blood osmolarity decreased (Investigations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results conducted at Site shall not be published before 1st multicenter publication by Sponsor but can proceed if there is no such publication ≤18 months after study completion/termination at all sites and all data have been received. Before submitting manuscript/materials to an outside person/entity, site shall give Sponsor 60 days to review and comment. Site shall, upon request, further delay publication/presentation for ≤120 days to allow Sponsor to protect its interests in Inventions.

DOCUMENTS (2):
  • Study Protocol (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT02713490/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT02713490/SAP_001.pdf